CLINICAL TRIAL: NCT06165861
Title: The Effect of the Use of Virtual Reality Glasses on Surgical Fear and Anxiety in Patients Before Open Heart Surgery
Brief Title: The Effect of Using Virtual Reality Glasses on Surgical Fear and Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trakya University (Other)
Responsible Party: Principal Investigator, Seher Ünver, Associate Professor, Trakya University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2021-GOBAEK-452
Record Dates: First submitted 2023-11-21; First posted 2023-12-12 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2023-12

CONDITIONS: Open Heart Surgery; Virtual Reality; Preoperative Anxiety; Fear; Nurse
Keywords: open heart surgery; virtual reality; preoperative anxiety; surgical fear; surgery nurse

STUDY DESIGN:
Intervention Model Description: The research will be conducted using randomized controlled, experimental type and single-blind research methods. For this purpose, after the data are collected, they will be coded as A and B groups, so the researcher who will make the research statistics will analyze the data without knowing the study and control groups. Randomization method will be used to determine the groups. For this, the patients who meet the study criteria and volunteer will be assigned to the groups using the randomization program 'Random Allocation Software 2.0' according to the order of hospitalization.
Who Masked: Outcomes Assessor
Masking Description: The data analyse is going to be completed by a independent researcher.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental (with VR-G) (Experimental): The patients in this procedure watched video with using VR-G for approximately 6 minutes at the surgical clinic before going surgery.
  Interventions: Other: Experimental (with VR-G)
- Standard (No VR-G) (No Intervention): The patients took the standart protocol of the surgical clinic and didn't watch video with using VR-G

INTERVENTIONS:
Other: Experimental (with VR-G) — Watching video with using VR-G before undergoing open heart surgery
  Arms: Experimental (with VR-G)

SUMMARY:
The purpose of this clinical study is to evaluate the effect of using virtual reality glasses on the surgical fear and anxiety levels of patients undergoing open heart surgery on the morning of surgery. The main hypotheses are:

1. The surgical fear level of patients who use virtual reality glasses on the morning of surgery is lower than patients who do not use virtual reality glasses.
2. The anxiety level of patients who use virtual reality glasses on the morning of surgery is lower than patients who do not use virtual reality glasses.

Before the surgery, study group patients will be asked to watch videos using virtual reality glasses.

DETAILED DESCRIPTION:
The group distribution of the patients was made using the Random Allocation Software (Version 2.0.0) program and the patients were divided into two groups: the study group and the control group.

Patients in the study group were asked to watch videos using virtual reality glasses between the first, second and third evaluation before surgery.

The researcher visited the patients in the cardiovascular surgery ward before the surgery and reported that the patients in the study group would watch video (including nature sounds such as bird sounds, water sounds, etc) with virtual reality glasses. Patients in the control group were informed that the normal service protocol would be applied.

The Surgical Fear Scale was developed to measure the surgical fear levels experienced by patients before surgery. To assess surgical fear, patients are asked to rate their fear level for each question with a number ranging from 0 - 'I am not afraid at all' to 10 -'I am very afraid'. Visual Analog Scale - To evaluate anxiety, patients are asked to mark the anxiety they perceive on a line ranging from 0 -'no anxiety' to 10 -'highest level of anxiety'. The total score of the surgical fear scale is obtained by summing the scores of all scale questions; The lowest score that can be obtained is 0 and the highest score is 80. A lower score indicates that patients experience less surgical fear during their activities. Higher scores indicate a higher level of surgical fear.

To perform the first evaluation in the study group, the researcher went to the patient and evaluated the patient introduction form and surgical fear and anxiety levels. Then, the researcher nurse explained that they were waiting for the operating room team to arrive and gave the patients brief information about the virtual reality glasses. Then, entrances and exits to the room were restricted to ensure that the room was quiet enough to watch videos and away from distracting elements. Patients were then asked to watch the video carefully and focus on the video sounds. Virtual reality glasses were fitted to the patients and videos were started to be watched. The nurse researcher remained in the patient's room until the video ended. At the end of the video, the glasses were taken from the patient and disinfected, and the researcher nurse left the patient room. Then, a second evaluation was made by the service nurse. The third evaluation was made by the researcher nurse when the patients were taken down to the operating room waiting room.

In the control group, the first evaluation was made by the researcher nurse. Then, normal service protocol was applied to the control group patients and a second evaluation was made by the service nurse before going down to the operating room waiting room. The third evaluation was made by the researcher nurse in the operating room waiting room.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the research,
* Will undergo open surgery,
* Will undergo planned surgical intervention,
* Being over 18 years of age,
* No visual impairment,
* No hearing impairment,
* No speech impediment,
* Lack of a psychiatric diagnosis was included.

Exclusion Criteria:

* Having an emergency surgical procedure
* Having a visual impairment
* Having a hearing impairment
* Being under 18 years of age
* Lack of mental health
* Having a speech impediment

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2022-02-14 (Actual); Primary Completion 2023-06-16 (Actual); Study Completion 2023-10-16 (Actual)

PRIMARY OUTCOMES:
Surgical Fear | one day
  • Surgical fear level [Time Frame: Measurements will start in the surgical ward in the morning of the surgery day before gowning the surgery clothes (such as surgical gown, caps) and will end in the waiting room before transferring to the operating room.]
  o It will be evaluated using the Surgical Fear Scale. To assess surgical fear, patients are asked to rate their fear level for each question with a number ranging from 0 - "I am not afraid at all" to 10 - "I am very afraid".
Surgical Anxiety | one day
  • Anxiety level [Time Frame: Measurements will start in the surgical ward in the morning of the surgery day before gowning the surgery clothes (such as surgical gown, caps) and will end in the waiting room before transferring to the operating room.]
  o It will be evaluated using the Visual Analog Scale-Anxiety Scale. To assess anxiety, patients are asked to mark their perceived anxiety level on a horizontal line ranging from 0 - "no anxiety" to 10 - "highest anxiety level".

CONTACTS AND LOCATIONS:
Overall Officials: Seher Ünver, Principal Investigator — Trakya University; Tuba Erol Akar, Principal Investigator — Trakya University
Locations (1):
- Seher Ünver, Edirne, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Erol Akar T, Unver S. Effectiveness of Virtual Reality Glasses on Surgical Fear and Anxiety in Patients Before Open-heart Surgery: A Double-blind Randomized Controlled Trial. J Perianesth Nurs. 2025 Jun;40(3):682-688. doi: 10.1016/j.jopan.2024.08.011. Epub 2024 Nov 30. PMID 39614857